CLINICAL TRIAL: NCT01389908
Title: A Follow up Study of Intramuscular Olanzapine Depot in Patients With Schizophrenia or Schizoaffective Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shalvata Mental Health Center (Other)
Responsible Party: Dr. Ziv Carmel, Shalvata MHC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: sh-03-11
Record Dates: First submitted 2011-06-30; First posted 2011-07-08 (Estimated); Last update posted 2011-07-08 (Estimated); Status verified 2011-06

CONDITIONS: Schizophrenia; Schizoaffective Disorders
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Olanzapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- schizophrenia (Experimental): schizophrenia or schizoaffective patients
  Interventions: Drug: olanzapine

INTERVENTIONS:
Drug: olanzapine — Patients will receive doses within the range of 280 mg to 405mg OP Depot, according the physician's judgment, on a 3-week interval.

SUMMARY:
The purpose of this study is to assess the long-term efficacy of Olanzapine Pamoate (OP) Depot in patients diagnosed with schizophrenia or schizoaffective disorder.

DETAILED DESCRIPTION:
Since its introduction in the United States and Europe in the mid-1990s, olanzapine has been distinguished from other antipsychotic medications (including other "atypical" compounds) by its superior efficacy and safety profiles (Beasley et al. 1996a, 1996b; Tollefson et al. 1997).

Only older "typical" antipsychotics have been available in long-acting (depot) formulations. They are most frequently prescribed to enhance compliance and, to a lesser degree, for convenience, as the need for daily oral dosing is eliminated. The popularity of depot formulations has diminished since the introduction of highly effective oral atypical antipsychotics with vastly reduced side effects. However, long-acting injections remain an important treatment option for many patients with psychotic disorders, and the need to provide a safer, more effective depot formulation to this population is compelling. Accordingly, an "atypical" depot of olanzapine, which can be administered every 2 to 4 weeks, has been developed to enhance convenience and compliance with antipsychotic therapy.

The depot formulation of olanzapine (LY170053) to be evaluated in this study is olanzapine pamoate monohydrate (OPM) (the salt of pamoic acid and olanzapine), suitable for deep intramuscular injection. Olanzapine Pamoate (OP) Depot (formerly referred to as IM olanzapine depot in previous versions of protocol) consists of OPM powder, which is suspended in an aqueous vehicle immediately prior to use. Several pamoate salts of other registered drug products are currently approved for chronic oral administration in the United States (for example, hydroxyzine pamoate and imipramine pamoate). Another pamoate salt depot for intramuscular injection has also been approved in the US (TrelstarTM LA, triptorelin pamoate for injectable suspension) for the treatment of prostate cancer.

As of March 2002, the pamoate formulation of OP Depot has been tested in 12 healthy subjects and approximately 250 patients with schizophrenia in 2 clinical pharmacology studies, F1D-EW-LOAZ and F1D-EW-LOBE, respectively, and one receptor occupancy (positron emission tomography) study, F1D-EW-HGJW. Dosages included single doses up to 450mg and multiple doses up to 405mg every 4weeks.

This open-label study will assess long-term efficacy 280 mg to 405mg of OP Depot administered on a 3-week interval in patients with schizophrenia or schizoaffective disorder

ELIGIBILITY:
Inclusion Criteria:

* Two patients that have been stabilized on OP Depot will be enrolled to the follow-up study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2011-06; Primary Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
blood pressure and pulse | 10 minutes prior to the injection
  supine and standing blood pressure and pulse will be measured 10 minutes prior to the injection
blood pressure and pulse | 15 minutes following the injection
  supine and standing blood pressure and pulse will be measured 15 minutes following the injection

CONTACTS AND LOCATIONS:
Locations (1):
- Shalvata MHC, Hod HaSharon, Israel